CLINICAL TRIAL: NCT01907516
Title: Managing Diabetes in Pregnancy Using Cell Phone/Internet Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawaii Pacific Health (Other)
Collaborators: Hawaii Medical Service Association (Other); Hookele Personal Health Planners (Unknown); Kapiolani Medical Center For Women & Children (Other)
Responsible Party: Principal Investigator, Marguerite Lisa Bartholomew, MD, Physician, Hawaii Pacific Health
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2009-118
Record Dates: First submitted 2013-07-22; First posted 2013-07-25 (Estimated); Results first posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes During Pregnancy; Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cell phone-internet first (Active Comparator): Cell phone-internet home glucose reporting system first
  Interventions: Device: Cell phone-internet home glucose reporting system; Behavioral: Voicemail home blood glucose reporting
- Voicemail first (Placebo Comparator): Voicemail home blood glucose reporting first
  Interventions: Device: Cell phone-internet home glucose reporting system; Behavioral: Voicemail home blood glucose reporting

INTERVENTIONS:
Device: Cell phone-internet home glucose reporting system — Glucose monitoring via cell phone and internet using the Confidant Diabetes Management Application and the Confidant Connector.
  Other Names: Confidant System
Behavioral: Voicemail home blood glucose reporting — Glucose monitoring via standard telephone and fax reporting.

SUMMARY:
To compare compliance and satisfaction between a traditional method of blood glucose reporting using voicemail (control) and a novel method using cell phone /internet (Confidant) technology in the management of diabetic pregnant women.

DETAILED DESCRIPTION:
Control of blood glucose levels is beneficial during pregnancy, however, the ability to effectively monitor patient's blood glucose levels is challenging and time consuming for patients and care providers. Patients must keep track of their own glucose levels and take the initiative to check blood glucose multiple times per day. Traditionally, patients record their glucose levels in a logbook, which they bring with them during an office visit or use to report their glucose levels over the phone. Non compliance and factitious reporting are not uncommon. Obstetricians and or diabetes program staff spend hours communicating with patients to obtain and record glucose values therefore alternatives to phone calls are needed.

Investigators performed a prospective randomized cross over study comparing a conventional voicemail (control) system for home glucose reporting with a cell phone/internet reporting system (Confidant). The primary outcome measure was compliance with home blood glucose fingerstick reporting. Compliance was determined by the number of home glucose fingersticks reported / expected (%). The secondary outcome was patient satisfaction. Subjects were participants in the Kapiolani Medical Center for Women and Children's diabetes in pregnancy program known as "A Sweeter Choice". IRB approval was obtained before starting the study and all subjects received informed consent. The study was funded by Hawai'i Medical Service Association, a medical insurance company in Hawaii. The Confidant equipment was supplied by Hookele Personal Health Planners, LLC. None of the Ho'okele or Hawaii Medical Service Association staff were involved in data collection or analysis. Study subjects were randomized to Confidant or the control system at the entry into the diabetes program during consultation with the Maternal Fetal Medicine physician. After randomization, subjects performed the assigned monitoring system for 3 weeks. After three weeks, they switched to the other monitoring system. A satisfaction survey was completed after three weeks on the second system was completed.

ELIGIBILITY:
Inclusion Criteria:

-Pregnant women >=18 years with gestational diabetes or pregestational Type 2 diabetes referred to the diabetes in pregnancy management program before 30 weeks 1 day gestation.

Exclusion Criteria:

* Age less than 18 year
* Pregnancy >=30 weeks 1 day
* Type I pregestational diabetes
* Inability to speak English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-02; Primary Completion 2010-08 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marguerite L Bartholomew, MD, Principal Investigator — John A Burns University of Hawaii School of Medicine
Locations (1):
- Kapiolani Medical Center for Women and Children, Honolulu, Hawaii, United States

REFERENCES:
- [Background] Jackson CL, Bolen S, Brancati FL, Batts-Turner ML, Gary TL. A systematic review of interactive computer-assisted technology in diabetes care. Interactive information technology in diabetes care. J Gen Intern Med. 2006 Feb;21(2):105-10. doi: 10.1111/j.1525-1497.2005.00310.x. Epub 2005 Dec 22. PMID 16390512

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were participants in the Kapiolani Medical Center for Women and Children's (KMCWC) diabetes in pregnancy program known as "A Sweeter Choice". Subjects were enrolled between February 4, 2009 and 3/11/2010.
Groups:
- Cell Phone-internet First, Then Voicemail: Cell phone-internet home glucose reporting system first, then voicemail
- Voicemail First, Then Cell Phone-internet: Voicemail home blood glucose reporting first, then cell phone-internet
Period: First Intervention (3 Weeks)
Arm/Group | Cell Phone-internet First, Then Voicemail | Voicemail First, Then Cell Phone-internet
Started | 50 | 50
Completed | 40 | 34
Not Completed | 10 | 16
Not completed — Withdrawal by Subject | 5 | 9
Not completed — Lost to Follow-up | 1 | 3
Not completed — Delivered before second arm | 3 | 4
Not completed — Developed DKA during study | 1 | 0
Period: Second Intervention (3 Weeks)
Arm/Group | Cell Phone-internet First, Then Voicemail | Voicemail First, Then Cell Phone-internet
Started | 40 | 34
Completed | 40 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cell Phone-internet First, the Voicemail: Cell phone-internet home glucose reporting system first
- Voicemail First, Then Cell Phone-internet: Voicemail home blood glucose reporting first
- Total: Total of all reporting groups
Arm/Group | Cell Phone-internet First, the Voicemail | Voicemail First, Then Cell Phone-internet | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.79 (4.94) | 32.5 (5.76) | 33.12 (5.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Compliance With Home Blood Glucose Reporting
Description: Compliance was calculated as a percentage for each method (Confidant or Voicemail) by dividing the total number of reported glucose readings among all participants by the total number of expected readings (4 daily) over the 6 week study time period. Women with gestational diabetes are instructed to monitor their glucose 4 times per day.
Time Frame: 6 weeks
Measure: Number; unit: percentage of expected glucose tests
Groups:
- Used Confidant Method: Cell phone-internet home based glucose monitoring first, then conventional Voicemail system for home glucose reporting
- Used Voicemail Method: Voicemail first, then cell phone-internet home glucose monitoring system
Arm/Group | Used Confidant Method | Used Voicemail Method
Number analyzed (Participants) | 74 | 74
percentage of expected glucose tests | 89.3 | 87.6

2. Secondary Outcome: Subject Satisfaction
Description: Satisfaction was measured with a survey after completing using both reporting methods
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Groups:
- Total Study Population: All study participants, includes those in cell phone-internet first, then voicemail and voicemail first, then cell phone-internet
Arm/Group | Total Study Population
Number analyzed (Participants) | 74
percentage of participants | 67

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Cell Phone-internet First, Then Voicemail: Cell phone-internet home glucose reporting system first
Arm/Group | Cell Phone-internet First, Then Voicemail | Voicemail First, Then Cell Phone-internet
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
Selection bias towards English speaking, educated, and technology savvy women, a 25% drop out rate, a high rate of glucose reporting compliance in the control system, and technical problems when Confidant first started which were quickly resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No